CLINICAL TRIAL: NCT05175482
Title: The Impact of Health Belief Model Based Education on Human Papilloma Virus Infection and Vaccination Among University Students: A Randomized Controlled Trial
Brief Title: Health Belief Model Based Education on Human Papilloma Virus Infection and Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Betul Okuyan, Assoc.Prof., Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MARCPD-002
Record Dates: First submitted 2021-12-12; First posted 2022-01-03 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Human Papilloma Virus; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education received group (Experimental): Health belief model based education on HPV infection and vaccination
  Interventions: Other: Virtual Education
- Control Group (No Intervention): No virtual education

INTERVENTIONS:
Other: Virtual Education — health belief model based virtual education
  Arms: Education received group

SUMMARY:
To evaluate impact of Health Belief Model Based Education on Human Papilloma Virus Infection and Vaccination among University Students

DETAILED DESCRIPTION:
In this randomized controlled study, it aims to evaluate impact of Health Belief Model based virtual education on Human Papilloma Virus Infection and Vaccination among University Students.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18 years or over

Exclusion Criteria:

* University students have been received HPV vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 127 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline assessment of knowledge level on Human Papilloma Virus (HPV) Infection and Vaccination at first day | baseline and next day after the education (at first day)
  The scale consists of 10 items. A higher score represents a higher knowledge level.
Change from baseline score of Human Papilloma Virus (HPV) Infection and Vaccination Health Belief Model Scale at first day | baseline and next day after the education (at first day)
  The scale consists of 14 items. The construction of the scale consists of perceived severity (n=4 items), perceived susceptibility (n=2 items), perceived benefit (n=3 items), perceived barriers (n=5 items). A 4-point Likert scale was used to assess each item.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Okuyan, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)